CLINICAL TRIAL: NCT06121037
Title: Greater Occipital Nerve Pulsed Radiofrequency for the Treatment of Combined Migraine and Cervicogenic Headache (New Approach): Randomized Clinical Trial
Brief Title: Greater Occipital Nerve Pulsed Radiofrequency for the Treatment of Combined Migraine and Cervicogenic Headache (New Approach)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Mohammed AboelFadl, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GON RF
Record Dates: First submitted 2023-11-02; First posted 2023-11-07 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Greater Occipital Nerve; Pulsed Radiofrequency

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proximal group (Experimental): proximal ultrasound-guided GON radiofrequency ablation
  Interventions: Procedure: proximal ultrasound-guided GON radiofrequency ablation
- Distal group (Experimental): distal ultrasound-guided GON radiofrequency ablation
  Interventions: Procedure: distal ultrasound-guided GON radiofrequency ablation

INTERVENTIONS:
Procedure: proximal ultrasound-guided GON radiofrequency ablation — proximal GON radiofrequency
  Arms: Proximal group
Procedure: distal ultrasound-guided GON radiofrequency ablation — distal GON radiofrequency
  Arms: Distal group

SUMMARY:
Combined migraine and cervicogenic headache present significant challenges in clinical management due to their complex and overlapping pathophysiologies. Both conditions involve the trigeminocervical complex, suggesting a potential shared anatomical and neurobiological basis

DETAILED DESCRIPTION:
Traditional treatment approaches for these headaches often include pharmacological interventions, but in cases of refractory or inadequate response, interventional techniques targeting the greater occipital nerve (GON) have gained attention.

Radiofrequency ablation (RFA) has gained recognition as a potential therapeutic option for patients with refractory combined migraine and cervicogenic headaches. The proximal and distal ultrasound-guided approaches are widely utilized for GON RFA. These approaches aim to disrupt pain signals transmitted by the GON and provide relief of pain for these headache disorders

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with combined migraine and cervicogenic headache according to The International Classification of Headache Disorders (ICHD)
* Age between 18 and 65 years.
* Willingness to participate and provide informed consent

Exclusion Criteria:

* Previous neurosurgical procedures for headache management.
* Patients with contraindications for the RF technique
* Pregnancy or lactation
* History of psychiatric disorders or substance abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Numerical rating score | baseline and at follow-up visits (2 weeks.1, 2.3, and 6 months)
  0-10 scale, with 0 indicating no pain and 10 indicating the worst possible pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut governorate, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Batistaki C, Madi AI, Karakosta A, Kostopanagiotou G, Arvaniti C. Pulsed Radiofrequency of the Occipital Nerves: Results of a Standardized Protocol on Chronic Headache Management. Anesth Pain Med. 2021 Oct 6;11(5):e112235. doi: 10.5812/aapm.112235. eCollection 2021 Oct. PMID 35075408
- [Background] Cohen SP, Peterlin BL, Fulton L, Neely ET, Kurihara C, Gupta A, Mali J, Fu DC, Jacobs MB, Plunkett AR, Verdun AJ, Stojanovic MP, Hanling S, Constantinescu O, White RL, McLean BC, Pasquina PF, Zhao Z. Randomized, double-blind, comparative-effectiveness study comparing pulsed radiofrequency to steroid injections for occipital neuralgia or migraine with occipital nerve tenderness. Pain. 2015 Dec;156(12):2585-2594. doi: 10.1097/j.pain.0000000000000373. PMID 26447705